CLINICAL TRIAL: NCT06748131
Title: Efficiency of Operating Room Simulation for Training Medical Students in the MEDI045 Program at King Saud University
Brief Title: Efficiency of Operating Room Simulation for Training Medical Students at King Saud University (EORMST-KSU)
Acronym: EORMST-KSU
Status: Active, not recruiting | Type: Observational
Sponsor: King Saud Medical City (Other Government)
Responsible Party: Principal Investigator, Walid Mohamed Ragab Mohamed Badwi, Resident anesthesia,MD,MBBCH,EDAIC PART1, King Saud Medical City
Other Study IDs: KingSaudMC; 2024;Ref. No. 24/1145/IRB (Other: IRB of the College of Medicine,KSU, Riyadh, SA)
Record Dates: First submitted 2024-12-16; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Operating Rooms; High Fidelity Simulation Training
Keywords: Operating room simulations; High fidelity simulation; Medical student training; Anesthesia education; Clinical decision-making

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate the effectiveness of operating room (OR) simulation-based training in improving anesthesia skills and decision-making for medical students at King Saud University. Specifically, the study focuses on the integration of SimMan 3G technology and high-fidelity simulation scenarios within the MEDI045 Basic Anesthesia and Resuscitation course.

By engaging in realistic, high-stress scenarios, the students will practice essential tasks such as airway management, anesthesia administration, and patient surveillance. The goal is to enhance students' technical skills, critical decision-making, and ability to adapt to dynamic clinical conditions.

In addition to evaluating improvements in anesthesia competencies, the study also seeks to assess student satisfaction and confidence levels after completing the simulation-based training. The research will contribute to a better understanding of how simulation can bridge the gap between theoretical knowledge and practical application in anesthesia education.

Data collected will include quantitative measures of technical proficiency and decision-making effectiveness, along with qualitative feedback regarding students' experiences, perceptions of competency, and overall satisfaction with the revised curriculum. The findings will help refine medical education practices, with a focus on patient safety, effective communication, and teamwork within the OR.

The study is being conducted at King Saud University and involves fourth-year medical students enrolled in the MEDI045 course.

DETAILED DESCRIPTION:
This study aims to assess the impact of simulation-based training on the development of anesthesia skills and clinical decision-making in medical students enrolled in the MEDI045 Basic Anesthesia and Resuscitation course at King Saud University. The primary intervention involves the integration of SimMan 3G high-fidelity simulators within the course curriculum, providing students with immersive, realistic scenarios that closely replicate the dynamic conditions of a real operating room (OR).

The key focus areas of the study include:

Technical Skills Development: The study will evaluate students' proficiency in performing essential anesthesia tasks, such as airway management, drug administration, and patient monitoring. Skills will be assessed through both pre- and post-simulation tests to measure improvements in technique and dexterity.

Decision-Making and Critical Thinking: By simulating high-pressure scenarios, the study aims to evaluate how well students make decisions under stress, particularly with respect to patient safety. Students' abilities to assess and respond to fluctuating clinical conditions will be analyzed, with a focus on minimizing errors and improving patient outcomes.

Student Adaptability: A key objective of the study is to measure students' adaptability in managing unforeseen complications. The simulations will expose students to a range of emergency situations, such as intraoperative crises, and evaluate their ability to maintain composure and provide effective care.

Student Satisfaction and Confidence: Post-simulation surveys and structured debriefing sessions will be used to gather qualitative data on student satisfaction and perceived confidence in their ability to manage anesthesia in real-world settings.

The study uses a mixed-methods research design, combining quantitative analysis (using pre- and post-test scores and statistical methods like t-tests and chi-square tests) with qualitative data (from surveys and debriefing sessions). The study will measure not only technical proficiency but also examine how simulation influences students' psychological readiness and communication skills within a team-based environment.

Data gathered will be used to evaluate the effectiveness of simulation-based training in improving both anesthesia skills and decision-making abilities. The results will inform future curriculum improvements, with the goal of enhancing patient safety, communication, and teamwork within medical education.

ELIGIBILITY:
Inclusion Criteria:

* Medical students enrolled in the MEDI045 Basic Anesthesia and Resuscitation course at King Saud University.
* Students in their fourth year of medical school.
* Consent to participate in simulation-based training and data collection.
* Ability to understand and follow instructions in English.

Exclusion Criteria:

* Students who have previously undergone simulation-based anesthesia training.
* Students who are not in good academic standing.
* Students with documented medical conditions that could affect their ability to participate in simulation sessions (e.g., severe anxiety or motion sickness).

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study will involve fourth-year medical students from the MEDI045 Basic Anesthesia and Resuscitation course at King Saud University, Riyadh, Saudi Arabia. These students will undergo simulation-based training designed to enhance their technical and decision-making skills in anesthesia. Students will be assessed for their proficiency and adaptability in anesthesia skills before and after participating in the simulation training sessions.
Sampling Method: Non-Probability Sample
Enrollment: 10911 (Estimated)
Dates: Start 2024-03-03 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-03-03 (Estimated)

PRIMARY OUTCOMES:
Change in Technical Anesthesia Skills Following Simulation-Based Training | Pre-training (baseline) Post-training (immediately following the final simulation session) Follow-up assessments at 1 month and 3 months post-training
  This outcome will assess the change in technical proficiency in anesthesia-related procedures following simulation-based training using high-fidelity SimMan 3G simulators. Key skills assessed will include airway management, anesthesia induction and monitoring, and postoperative care. The assessment will be conducted at baseline (pre-training) and post-training (immediately following the final simulation session), with follow-up assessments at 1 month and 3 months to evaluate skill retention. The measurement tool used will be a skills assessment rubric specific to each procedure, with scores reflecting proficiency in each skill.

CONTACTS AND LOCATIONS:
Locations (1):
- King Saud University Medical City (KSUMC), College of Medicine, Riyadh, Saudi Arabia